CLINICAL TRIAL: NCT02620605
Title: The Influence of Timing of Cabergoline Initiation on Prevention of Ovarian Hyper Stimulation Syndrome in Patients Undergoing Intra Cytoplasmic Sperm Injection .
Brief Title: The Influence of Timing of Cabergoline Initiation on Prevention of OHSS
Acronym: OHSS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mona M Shaban (Other)
Responsible Party: Sponsor-Investigator, Mona M Shaban, Mona Mohamed shaban ,assistant professor MD, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: C123
Record Dates: First submitted 2015-11-24; First posted 2015-12-03 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Ovarian Hyperstimulation Syndrome
Keywords: Cabergoline; Ovarian Hyper Stimulation Syndrome (OHSS)
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome | interventions — Cabergoline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Late administration of Cabirgoline 0.5 mg (Active Comparator): Cabergoline 0.5mg (Dostinex®, Pfizer Australia Pty Ltd ) administrated once daily started on day of HCG triggering and continued for 8 days.
  Interventions: Drug: Late Cabergoline 0.5mg
- Early administration of Cabirgoline 0.5mg (Experimental): Cabergoline 0.5mg(Dostinex®, Pfizer Australia Pty Ltd ) once daily stared once patients fulfilling the inclusion criteria at any day of cycle and continued for 8 days post HCG trigger.
  Interventions: Drug: Early Cabergoline 0.5mg

INTERVENTIONS:
Drug: Late Cabergoline 0.5mg — Cabergoline 0.5mg will be administrated once daily at day of HCG trigger and continued for 8days
  Other Names: Dostenix (Dostinex®, Pfizer Australia Pty Ltd )
  Arms: Late administration of Cabirgoline 0.5 mg
Drug: Early Cabergoline 0.5mg — Cabergoline 0.5mg will be administrated once daily when E2 is more than 4000pg/ml and /or more than 18 follicles of 11mm diameter or more are encountered at any day of the controlled ovarian hyper-stimulation and before HCG trigger to be continued for 8days after HCG trigger.
  Other Names: Dostinex (Dostinex®, Pfizer Australia Pty Ltd )
  Arms: Early administration of Cabirgoline 0.5mg

SUMMARY:
Study the effect of early cabergoline administration in prevention of occurrence or decreasing the severity of OHSS in patients undergoing intra cytoplasmic sperm injection.And its effect on oocyte maturation,fertilization and pregnancy rate..

DETAILED DESCRIPTION:
Patients less than 35years undergoing Intra Cytoplasmic Sperm Injection for infertility scheduled for gonadotropin releasing hormone agonist long protocol of ovarian stimulation.

All patient will receive combined oral contraceptive pills (Gynera, Schering-plow: plough) starting from day 5 of cycle that precedes the stimulated cycle .On day 21 of that cycle all patients will start to receive Gonadotrophin releasing hormone agonist in the form of (decapeptyl 0.1 sc daily and continued till the day of HCG administration).

To ensure that all patients are completely down regulated and desensitized ,trans-vaginal ultrasound will be performed at day 2-3 of menses of stimulated cycle to ensure endometrial thickness less than 5 mm and no ovarian cysts.Also serum E2 level is less than 50 pg/ml.

Then all patients will start to receive Gonadotrophin ( HMG) (Menogon, ferring pharmaceuticals, Germany) 225 IU (international unit) Intramuscular Injection daily,with continuous scheduled follow up of ovarian response by serial trans -vaginal US to assess follicular growth together will serial serum E2 starting from day 6 of cycle and onwards.With adjustments of gonadotropin dose and monitoring frequency based on patient response.

During follow up once the recruited patients fulfilling the inclusion criteria (serum E2 equal or more than 4000 pg/ml and /or 18 or more follicles of 11 mm diameter or more at any day of stimulation),they will be allocated randomly by computer generated cards and assigned by sealed envelopes by the treating doctor at the outpatient clinic.

Group A : will receive cabergoline 0.5 mg/day for 8 days, starting in the day of HCG (human chorionic gonadotropin ) injection.

Group B: will receive cabergoline 0.5 mg/day once the criteria of inclusion criteria is fulfilled and continued till the day of human chorionic gonadotropin (HCG ) trigger and continued 8 days more from day of trigger .

ELIGIBILITY:
Inclusion Criteria:

* Female less than 35 years under going Intra cytoplasmic sperm injection cycle for infertility (tubal factor or un explained infertility).
* 18 or more oocyte 11 mm in diameter and/or E2 is more than 4000 pg/ml at any day of the stimulation cycle before or at HCG trigger

Exclusion Criteria:

* patient with one ovary
* patients already receiving cabergoline treatment
* Severe Male factor infertility.
* Thyroid dysfunction.

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2017-12-20 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Occurrence and severity of OHSS | 2 to 4weeks after trigger
  either early or late OHSS (early OHSS is the occurrence within 9 days after OPU and occurrence after 10 days was classified as late OHSS.The severity of OHSS was graded according to the criteria of Navot et al. (1992). Moderate OHSS in particular is characterized by abdominal distension and discomfort, nausea±vomiting±diarrhoea, enlarged ovaries 5-12 cm and ultrasonographic evidence of ascites. Severe OHSS is characterized by variable ovarian enlargement; massive ascites±hydrothorax; breathing difficulties; haematocrit >45%; white blood cell count >15 000; oligouria; creatinine 1.0-1.5;liver dysfunction; and anasarca oedema.)

SECONDARY OUTCOMES:
Number of M|| oocytes. | maximum one day after ovum pick up
Fertilization rate. | 16 to 19 hours after ICSI
  fertilization rate (the presence of two pronuclei (2PN) at the time of fertilization assessment, 16 to 19 hours after ICSI),
Clinical Pregnancy rate | 2 to 4 weeks after positive pregnancy test
  Clinical pregnancy was considered to be the presence of a gestational sac with fetal heart activity.
implantation rate | 2 to 4 weeks after positive pregnancy test
  implantation rate( the percentage of embryos which successfully undergo implantation compared to the number of embryos transferred)

CONTACTS AND LOCATIONS:
Overall Officials: Mona M Shaban, MD, Principal Investigator
Locations (1):
- IVF department in Kasr Alaini hospital,private IVF centre, Cairo, Egypt